CLINICAL TRIAL: NCT03163290
Title: Effect of Two Strengthening Protocols for Lower Limbs in Patients With Patellofemoral Pain: Randomized Clinical Trial
Brief Title: Effect of Two Strengthening Protocols for Lower Limbs in Patients With Patellofemoral Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Ceara (Other)
Responsible Party: Principal Investigator, Gabriel Peixoto Leão Almeida, Professor, Universidade Federal do Ceara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TCC_LARISSA NEVES
Record Dates: First submitted 2017-05-19; First posted 2017-05-23 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Posterolateral Hip Complex Exercises (Experimental): The intervention protocol will be composed of: Heating, lower limb stretching, strengthening the quadriceps, and hip abductors, lateral rotators and extensors. Posterolateral Hip Complex Exercises add extension knee in open kinetic chain, squat , abduction exercise, Clam exercise and external rotation exercise. Physiotherapy treatment sessions will last for an average of one hour, twice a week, for a period of six weeks.
  Interventions: Other: Posterolateral Hip Complex Exercises
- Anteromedial Hip Complex Exercises (Active Comparator): The intervention protocol will be composed of: Heating, lower limb stretching, strengthening the quadriceps, and hip aductors, medial rotators and flexors. Anteromedial Hip Complex Exercises add extension knee in open kinetic chain, squat ,hip adduction exercise, adduction with a ring between the thighs and internal rotation exercise. Physiotherapy treatment sessions will last for an average of one hour, twice a week, for a period of six weeks.
  Interventions: Other: Anteromedial Hip Complex Exercises

INTERVENTIONS:
Other: Posterolateral Hip Complex Exercises — The treatment protocol was composed of: Heating, lower limb stretching, strengthening the quadriceps e hip muscles. The following exercises were included: abduction exercise, Clam exercise and external rotation exercise
  Arms: Posterolateral Hip Complex Exercises
Other: Anteromedial Hip Complex Exercises — The treatment protocol was composed of: Heating, lower limb stretching, strengthening the quadriceps e hip muscles. The following exercises were included: hip adduction exercise, adduction with a ring between the thighs and internal rotation exercise.
  Arms: Anteromedial Hip Complex Exercises

SUMMARY:
Patellofemoral Pain (PFP) is one of the most common disorders that affecting the physically active population, and its incidence is higher among women. Despite the high incidence, the etiologies of this painful syndrome are still unclear. Research has verified the influence of hip stabilizers on knee injurie and has demonstrated a deficit of strength of the hip lateral rotator, abductors and extensors muscles in patients with PFP. The aim of this study is to compare the effectiveness of strengthening the Posterolateral Hip Complex with the Anteromedial Hip Complex associated with quadriceps strengthening for pain reduction and improvement of functional capacity in patients with PFP.

DETAILED DESCRIPTION:
The physical therapy sessions will average duration of one hour, often twice a week for six weeks. The exercise intensity will be monitored by the physiotherapist as determined by the participant's ability to complete 10 repetitions for a particular exercise and its difficulty of execution perceived by the modified Borg scale (CR-10). The exercises are performed with load between 60-80% of their capacity, the load will be increased from 2 to 10% when the patient can perform 14 full repetitions in the last series. It will be set to 30 seconds of rest between reps and 2 minutes between sets of exercise.

Both groups will perform prior heating exercises bike for 5 minutes with moderate intensity with the Borg scale. Then there will be one stretche repetitions held for 45 seconds of muscle groups: hamstrings, quadriceps, abductors, adductors and gastrocnemius. Thus, they will be performed strengthening exercises in extension and knee in open kinetic chain and squat.

The Posterolateral Hip Complex (PLC) add hip abduction exercise, Clam exercise and external rotation exercise. Studies prior point out that these exercises are among those withhigher electromyographic activity of the gluteus medius and maximus muscles.

The Anteromedial Hip Complex (AMC) add hip adduction exercise, adduction with a ring between the thighs and internal rotation exercise.

The exercises will be carried out to load 60-80% of 1 repetition maximum 8-12 reps, 1-3 sets and 2-3 times a week. All exercises are performed without worsening pain and intensity of exercise will be controlled according to the perceived exertion scale of Borg.

ELIGIBILITY:
Inclusion Criteria:

* Practicing physical activity for at least 3 times a week for at least 30 minutes;
* Pain localized specifically around the patellofemoral joint, pain reproduced or reported in at least two of the following criteria: up or down stairs, squatting, kneeling, sitting for a long time, isometric contraction of the quadriceps, jumping, running and pain on palpation of the lateral and / or medial facet of the patella;
* Report pain of insidious onset and lasting at least three months;
* Pain at least three in the Numerical Pain Scale during the last week;
* Report a maximum of 86 points on the Anterior Knee Pain Scale (maximum = 100 points).

Exclusion Criteria:

* Previous surgery on the hip, knee, ankle and / or spine;
* History of patellar dislocation;
* Clinical evidence of knee instability (anterior and posterior drawer test, Lachman, varus and valgus stress);
* Meniscal lesions or intra-articular lesions;
* Evidence of edema;
* Osgood-Schlatter syndrome or Sinding-Larsen-Johansson;
* Patellar tendinopathy;
* Chondral lesion;
* Osteoarthritis;
* Muscle or joint injuries to the hip.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2017-11-12 (Actual); Study Completion 2019-03-12 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Scale | Six weeks
  Pain was assessed by use of an 11-point Numeric Pain Scale, where 0 corresponded to no pain and 10 corresponded to worst imaginable pain.
  to worst imaginable pain.
Anterior Knee Pain Scale | Six weeks
  Anterior Knee Pain Scale assesses functional capacity and pain level during functional and specific activities for patients with PFP. This scale was translated and culturally adapted to the Brazilian Portuguese language,10 and the score ranges from 0 (worst) to 100 (best).

SECONDARY OUTCOMES:
Numeric Pain Scale | Six months
  Pain was assessed by use of an 11-point Numeric Pain Scale, where 0 corresponded to no pain and 10 corresponded to worst imaginable pain.
  to worst imaginable pain.
Anterior Knee Pain Scale | Six months
  Anterior Knee Pain Scale assesses functional capacity and pain level during functional and specific activities for patients with PFP. This scale was translated and culturally adapted to the Brazilian Portuguese language,10 and the score ranges from 0 (worst) to 100 (best).
Numeric Pain Scale on Step Down Test | Six weeks
  Pain was assessed by use of an 11-point Numeric Pain Scale on Step Down Test, where 0 corresponded to no pain and 10 corresponded to worst imaginable pain.
  to worst imaginable pain.
Dynamic Knee Valgus on Frontal Plane Projection Angle | Six weeks
  The dynamic knee valgus was assessed by the FPPA during the forward step-down test filmed with a digital camera (60 fps). FPPA was measured by the angle formed by the intersection of the lines between the anterior superior iliac spine and the center of the malleoli at the center of the femoral condyles. The step height was normalized to 10% of the height of each participant. All participants performed two training tests and three valid tests, with a five-second cadence for each test. The FPPA was calculated at the time of the heel touch on the ground by the Kinovea® Video Editor program. We considered a positive value as dynamic valgus and a negative value as dynamic varus.
Global Effect Perception Scale | Six weeks
  This scale has 11 points ranging from minus five points (extremely worse), Zero (no change) to five points (fully recovered). For all measures of perceived global effect the participants will be asked: "compared to the beginning of this episode, how would you describe your knee these days?" Positive scores represent better recovery and negative scores indicate worsening of symptoms.
Global Effect Perception Scale | Six months
  This scale has 11 points ranging from minus five points (extremely worse), Zero (no change) to five points (fully recovered). For all measures of perceived global effect the participants will be asked: "compared to the beginning of this episode, how would you describe your knee these days?" Positive scores represent better recovery and negative scores indicate worsening of symptoms.
Muscle strength | Six weeks
  Muscle strength of the hip abductors, adductors, lateral rotators and medial rotators will be assessed with a manual dynamometer (Nicholas Manual MuscleTester, Lafayette Instrument Company, Lafayette, Indiana, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel PL Almeida, MSc, Principal Investigator — Universidade Federal do Ceara
Locations (1):
- Federal University of Ceara, Fortaleza, Ceará, Brazil

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared.